CLINICAL TRIAL: NCT02589366
Title: A Phase I, Prospective, Open-Label, Comparison Study of Lymphoseek® and Vital Blue Dye as Lymphoid Tissue Targeting Agents in Patients With Known Cancer of the the Endometrium Who Are Undergoing Lymph Node Dissection
Brief Title: Lymphoseek as Lymphoid Tissue Targeting Agent in Patients With Cancer of the Endometrium
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Cardinal Health 414, LLC (Industry)
Responsible Party: Principal Investigator, Michael McHale, Associate Physician Diplomate, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRPP #141163
Record Dates: First submitted 2015-10-20; First posted 2015-10-28 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Endometrial Cancer
Keywords: Lymphoseek; endometrial cancer; sentinel lymph node; lymph node dissection
MeSH Terms: conditions — Endometrial Neoplasms | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran; Technetium; iso-sulfan blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lymphoseek plus Vital Blue Dye (Experimental): Lymphoseek plus Vital Blue Dye: Single dose of 50 µg Lymphoseek radiolabeled with 75 MBq Tc 99m injected pre-operatively followed by next day intra-operative administration of vital blue dye.
  Interventions: Drug: Lymphoseek plus Vital Blue Dye

INTERVENTIONS:
Drug: Lymphoseek plus Vital Blue Dye — intrapatient comparison of Lymphoseek with Vital Blue Dye in detecting lymph node metastases
  Other Names: Technetium TC 99M; Tilmanocept; Lymphazurin

SUMMARY:
Part of standard treatment for endometrial cancer is to remove one or more groups of lymph nodes (lymph node dissection). Lymph nodes are small, bean-shaped organs located within the body throughout the lymphatic system (the tissues and organs involved in immunity, which aids in the fight against infection and cancer).

The purpose of this study is to compare the safety and ability of Lymphoseek and a Vital Blue Dye (tracing agent) to find lymph nodes that may carry cancer from the tumor through the lymphatic system. Lymphoseek will be injected into the tumor on the day before surgery to remove lymph nodes. Vital Blue Dye will be administered during surgery to trace the cancer as well. The surgeon will remove the lymph nodes as part of routine surgery and will keep track of which lymph nodes are identified by Lymphoseek and Vital Blue Dye. These nodes will be sent to another doctor to view them under a microscope and see if the nodes contain cancer cells.

The hypothesis is that Lymphoseek can be used safely and will be at least as effective as blue dye in identifying the lymph nodes that may have cancer cells.

DETAILED DESCRIPTION:
This is an open-label, single center, intra-patient safety and comparison study of Lymphoseek (Technetium Tc 99m Tilmanocept) and vital blue dye for the detection of lymph nodes in patients with endometrial cancer that are undergoing a lymph node dissection as part of their standard medical care.

The day before surgery, patients will have their tumor injected with 50 µg Lymphoseek radiolabeled with 75 megabecquerel (MBq) Tc 99m. Vital signs will be monitored for thirty minutes and then patients will undergo a whole body scan and single photon emission computed tomography/ x-ray computed tomography (SPECT/CT) one to two hours after Lymphoseek injection.

Fourteen to twenty hours after injection of Lymphoseek, patients will have a physical exam and clinical laboratory tests assessed prior to undergoing surgery. Sentinel lymph node identification begins with injection of Vital Blue Dye. Surgical access will be made to the lymphatic basins where nodes are expected to be. Sentinel lymph nodes will be identified by a hand-held gamma counter and/or blue appearance. The threshold criterion for positive "hot" nodes based on radioactivity is a count greater than the quantity of 3 square roots of the mean background count (i.e., standard deviation) added to the mean background count (referred to as the "3σ rule"). Once a lymph node has been identified, in vivo counts should be taken prior to excision. In vivo counts will consist of a set of three 1-second counts over the lymph node. A positive finding (i.e., localization) is a designated "hot" node (described above). Any lymph node count not meeting this threshold criterion will be considered a negative (non-localized) finding. To confirm the in vivo procedure, a set of three 1-second counts will be recorded for the excised lymph nodes. The count of the ex vivo lymph nodes will be compared to the room background counts, and the threshold criterion used to determine a positive finding for the in vivo nodes will be applied to the ex vivo specimens.

A thorough evaluation of the remaining lymphatic basin will be complete when all selected node counts are negative by use of the threshold criterion. The surgeon will continue with visualization and palpation according to local practice to ensure that no grossly positive lymph nodes remain at the site of resection. After identifying the sentinel lymph nodes, standard lymph node dissection will be performed. All removed lymph nodes are sent to pathology for further evaluation. All removed lymph nodes will be sent to pathology and will be confirmed for radioactive status (due to Lymphoseek) and blue appearance (due to vital blue dye. The pathological evaluation of lymph node(s) will include serial sectioning with H&E staining as well as immuno-histochemistry (IHC) stain according to institutional practice.

Patients will return for a routine post-operative follow-up visit 7-14 days after surgery for assessment of adverse events.

The primary objective is safety of Lymphoseek as measured by the incidence of adverse events, changes in laboratory values, vital signs and physical exam findings, and the radiation absorbed dose. Secondary evaluations include (1) the number of lymph nodes detected as "hot" by preoperative imaging (whole body scan and SPECT/CT) and intraoperative gamma detection, and (2) the rate of concordance between Lymphoseek and Vital Blue Dye in the in vivo detection of excised lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has provided written informed consent with Health Insurance Portability and Accountability Act (HIPAA) authorization.
2. The patient has diagnosed cancer of the endometrium.
3. The patient is a candidate for surgical intervention, with lymph node dissection being a part of the surgical plan.
4. The patient is at least 18 years of age at the time of consent.
5. The patient has an Eastern Cooperative Group (ECOG) performance status of Grade 0 - 2.
6. The patient has a clinical negative node status at the time of study entry (i.e., Tis-4, N0, M0).
7. If of childbearing potential, the patient has a negative pregnancy test within 72 hours before administration of Lymphoseek, has been surgically sterilized, or has been postmenopausal for at least 1 year.

Exclusion Criteria:

1. The patient is pregnant or lactating.
2. The patient has clinical or radiological evidence of metastatic cancer including palpably abnormal or enlarged lymph nodes (i.e., all patients should be any T, N0, M0).
3. The patient has a known hypersensitivity to Lymphazurin or Lymphoseek.
4. The patient has participated in another investigational drug study within 30 days of scheduled surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-11; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 0-15 days Postoperatively
  Adverse events experienced by the participants and radiation absorbed dose of injected Lymphoseek.

SECONDARY OUTCOMES:
Number of Lymphoseek positive lymph nodes detected preoperatively and intraoperatively. | 2 days
  Determination of the number of lymph nodes detected with Lymphoseek by preoperative whole body scan and SPECT/CT imaging and by intraoperative laparoscopic hand held gamma detection device
Number of lymph nodes identified intraoperatively as assessed by visualization and handheld gamma probe detection | 2 days
  Concordance of intraoperative detection rates of Lymphoseek and vital blue dye in histological evaluation and ultrastaging of resected lymph nodes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael McHale, MD, FACS, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No